CLINICAL TRIAL: NCT02677454
Title: Evaluation of a Flash Glucose Monitoring System in Ambulatory Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Libre
Record Dates: First submitted 2016-01-07; First posted 2016-02-09 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus
Keywords: Blood Glucose; Blood Glucose Self-Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flash Glucose Monitor (Experimental): Each patient with Type 1 diabetes will have a subcutaneous tissue FGM sensor inserted. The sensor will produce a maximum of 1440 tissue fluid glucose measurements per 24 hours and 20160 measurements during the 14 day study. The FGM data (Abbott Freestyle Libre) will be compared to the time-matched reference blood glucose measurements.
  Each ambulatory patient will sample capillary blood with the HemoCue meter and measure the concentration of glucose 6 to 10 times per day for 14 days. The concentration of finger-stick capillary blood glucose will be measured using the self-monitoring blood glucose (SMBG) hemocue meter in their daily living. The subjects will record SMBG, in a written diary. Subjects will dose insulin according to their routine methods throughout the 14 day study.
  Interventions: Device: Flash Glucose Monitor

INTERVENTIONS:
Device: Flash Glucose Monitor
  Other Names: Abbott Freestyle Libre

SUMMARY:
To evaluate the accuracy of the Flash Glucose Monitoring system (FGM), Abbot FreeStyle Libre, used today in clinical practice in Sweden in estimating plasma glucose levels. Data will be collected in ambulatory patients with type 1 diabetes to determine safety, accuracy, and reliability.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes
2. Adult patients, age 18 or older and < 75 years
3. Written informed consent -

Exclusion Criteria:

1. Pregnancy
2. Patients with severe cognitive dysfunction or other disease which makes FGM use difficult
3. History of allergic reaction to any of the FGMs materials or adhesives in Contact with the skin.
4. History of allergic reaction to chlorhexidine or alcohol anti-septic solution.
5. Continous Glucose Monitor (CGM) or FGM usage in the last month
6. Abnormal skin at the anticipated glucose sensor attachment sites(excessive hair, burn, inflammation, infection, rash, and/or tattoo)

   -

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Mean Absolute Relative Difference (MARD) | the whole study period, day 1-14
  Mean absolute relative difference (MARD) of all estimated capillary glucose values registered during the whole study period of the Freestyle Libre system compared to the capillary reference blood glucose measured with HemoCue.

SECONDARY OUTCOMES:
Mean absolute Difference (MAD) | the whole study period, day 1-14
  Mean absolute difference(MAD) of all estimated capillary glucose values registered during the whole study period of the Freestyle Libre System compared to the capillary reference blood glucose measured with HemoCue
Pearson Correlation Coefficient | the whole study period, day 1-14
  Pearson correlation coefficient (all values registered during the whole study period)between Freestyle Libre System compared to the capillary reference blood glucose measured with HemoCue
Mean absolute relative difference (MARD) | the whole study period, day 1-14
  The MARD registered during day 1-7 and day 8-14 separately of the Freestyle Libre system compared to the capillary reference blood glucose measured with HemoCue
Mean absolute difference MAD | the whole study period, day 1-14
  The MAD registered during day 1-7 and day 8-14 separately of the Freestyle Libre system compared to the capillary reference blood glucose measured with HemoCue
Pearson Correlation | the whole study period, day 1-14
  The Pearson Correlation (data registered during day 1-7 and day 8-14 separately) between Freestyle Libre system compared to the capillary reference blood glucose measured with HemoCue
Mean absolute relative difference (MARD) | the whole study period, day 1-14
  The MARD,(for data registered inte the following specified glucose ranges: < 4mmol/l, 4-10mmol/l and >10mmol/l) durin the whole study period of the Freestyle Libre system compared to the capillary reference blood glucose measured the HemoCue
Mean absolute difference (MAD) | the whole study period, day 1-14
  The MAD,(for data registered inte the following specified glucose ranges: < 4mmol/l, 4-10mmol/l and >10mmol/l) durin the whole study period of the Freestyle Libre system compared to the capillary reference blood glucose measured the HemoCue
Pearson Correlation | the whole study period, day 1-14
  The Pearson Correlation (for data registered inte the following specified glucose ranges: < 4mmol/l, 4-10mmol/l and >10mmol/l) between Freestyle Libre system compared to the capillary reference blood glucose measured with HemoCue
questionnaire | the whole study period, day 1-14
  The evaluation of the Freestyle Libre system from a questionnaires rated on a VAS-scale (Visual analogue scale), lowest value (0) equaling to Not true at all and highest value (10) equaling to Completely true

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Lind, MD, Phd, Principal Investigator — NU-Hospital Organization, Sweden
Locations (1):
- NU-Hospital Group, Uddevalla, Sweden

IPD SHARING:
Plan to Share IPD: No